CLINICAL TRIAL: NCT02730403
Title: Treatment-as-Usual (TAU) Opioid Use Outcomes Following Discharge From Detoxification and Short Term Residential Programs Affiliated With National Institute on Drug Abuse (NIDA) CTN-0051
Brief Title: TAU Opioid Use Outcomes Following Discharge From Detoxification and Short Term Residential Programs Affiliated With CTN-0051
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 16-00090
Record Dates: First submitted 2016-03-21; First posted 2016-04-06 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Opioid Use Disorder Patients
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Other: Treatment As Usual

SUMMARY:
This is an observational, "ancillary study" intended to describe opioid use among opioid use disorder patients following their discharge into the community from inpatient detoxification and/or short-term residential treatment programs affiliated with parent study CTN-0051, which assessed the comparative effectiveness of extended release injectable naltrexone (XR-NTX, Vivitrol®), an opioid antagonist recently approved and indicated for the prevention of relapse to opioid dependence, versus buprenorphine-naloxone (BUP-NX, Suboxone®), a high affinity partial agonist indicated for maintenance treatment of opioid dependence, as pharmacotherapeutic aids to recovery.

DETAILED DESCRIPTION:
Participant recruitment will begin after recruitment for CTN-0051 has been completed. Opioid use disorder patients will be recruited prior to leaving detoxification and/or short-term residential programs. Screening and baseline data (focused on demographics, diagnosis and service utilization) will be collected prior to discharge, and follow-up data (focused on opioid use) will be collected at weeks 1, 4 and 8 following discharge.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* Meet DSM-5 criteria for opioid-use disorder (heroin or prescription opioids);
* Have used opioids other than as specifically prescribed within thirty days prior to consent
* Seeking treatment for opioid dependence;
* Able to provide written informed consent;
* Able to speak English sufficiently to understand the study procedures.

Exclusion Criteria:

* Serious medical, psychiatric or substance use disorder that, in the opinion of the Site PI, would make participation hazardous to the participant, compromise study findings or prevent the participant from completing the study;
* Suicidal or homicidal ideation that requires immediate attention;
* Maintenance on methadone at doses of 30mg or greater at the time of signing consent;
* Presence of pain of sufficient severity as to require ongoing pain management with opioids;
* Pending legal action or other reasons that might prevent an individual from completing the study;
* If female, currently pregnant or breastfeeding or planning on conception;
* Prior participation in parent trial CTN-0051

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be a convenience sample of up to three hundred sixty (360) opioid dependent patients leaving detoxification or short-term residential units at sites participating in CTN-0051. Up to 60 participants will be recruited at each of approximately six sites.
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Rotrosen, MD, Principal Investigator — New York University Medical School
Locations (5):
- United States (5):
  - Tarzana Treatment Centers, Tarzana, California
  - Gateway Community Services, Inc., Jacksonville, Florida
  - Stanley Street Treatment and Resources, Fall River, Massachusetts
  - Bellevue Hospital, New York, New York
  - Maryhaven, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment As Usual: Patients admitted to detoxification or short term residential programs associated with CTN-0051 for Opioid Use Disorder (OUD).
Period: Overall Study
Arm/Group | Treatment As Usual
Started | 211
Completed | 157
Not Completed | 54

BASELINE CHARACTERISTICS:
Groups:
- Treatment As Usual: Patients admitted to detoxification or short term residential programs associated with CTN-0051 with OUD.
Arm/Group | Treatment As Usual
Number analyzed (Participants) | 211
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 211
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (9.48)
Age, Customized [Count of Participants; unit: Participants]
  18 - <25 | 23
  25 - <35 | 96
  35 - <45 | 52
  45 - <55 | 33
  55 - <65 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 156
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37
  Not Hispanic or Latino | 172
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 4
  Race: Asian | 1
  Race: Native Hawaiian or Other Pacific Islander | 1
  Race: Black or African American | 28
  Race: White | 143
  Race: More than one race | 10
  Race: Unknown or Not Reported | 24
Region of Enrollment [Number; unit: participants]
  United States | 211
Baseline Opioid Severity [Count of Participants; unit: Participants]
  Low | 110
  High | 101

OUTCOME MEASURES:

1. Primary Outcome: Days of Opioid Use
Description: Days of use during the first 4 weeks post discharge
Time Frame: Up to Week 4 Post Discharge
Measure: Mean (Standard Deviation); unit: days
Groups:
- Treatment As Usual: Patients admitted to detoxification or short term residential associated with CTN-0051 for OUD.
Arm/Group | Treatment As Usual
Number analyzed (Participants) | 211
days | 6.8 (8.95)

2. Primary Outcome: Positive Urine Drug Screen (UDS) at Week 1
Description: Number of positive UDSs at Week 1
Time Frame: week 1
Measure: Count of Participants; unit: Participants
Groups:
- Treatment As Usual: Patients admitted to detoxification or short term residential treatment programs associated with CTN-0051 with OUD.
Arm/Group | Treatment As Usual
Number analyzed (Participants) | 211
Participants | 106

3. Primary Outcome: Negative UDSs at Week 1
Description: Number of negative UDSs at Week 1
Time Frame: week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment As Usual
Number analyzed (Participants) | 211
Participants | 60

4. Primary Outcome: Missing UDSs at Week 1
Description: Number of missing UDSs at Week 1
Time Frame: week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment As Usual
Number analyzed (Participants) | 211
Participants | 45

5. Primary Outcome: Missing UDSs at Week 4
Description: Number of missing UDSs at Week 4
Time Frame: week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment As Usual
Number analyzed (Participants) | 211
Participants | 54

6. Primary Outcome: Positive UDSs at Week 4
Description: Number of positive UDSs at Week 4
Time Frame: week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment As Usual
Number analyzed (Participants) | 211
Participants | 102

7. Primary Outcome: Negative UDSs at Week 4
Description: Number of negative UDSs at Week 4
Time Frame: week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment As Usual
Number analyzed (Participants) | 211
Participants | 55

8. Primary Outcome: Missing UDSs at Week 8
Description: Number of missing UDSs at Week 8
Time Frame: week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment As Usual
Number analyzed (Participants) | 211
Participants | 55

9. Primary Outcome: Negative UDSs at Week 8
Description: Number of negative UDSs at Week 8
Time Frame: week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment As Usual
Number analyzed (Participants) | 211
Participants | 66

10. Primary Outcome: Positive UDSs at Week 8
Description: Number of positive UDSs at Week 8
Time Frame: week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment As Usual
Number analyzed (Participants) | 211
Participants | 90

11. Primary Outcome: Time to First Use
Description: Days to first opioid use from Timeline Followback
Time Frame: Up to Week 8 Post Discharge
Population: Patients admitted to detoxification or short term residential programs associated with CTN-0051 for OUD
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment As Usual
Number analyzed (Participants) | 211
days | 7.5 (10.17)

12. Primary Outcome: Time to Regular Use
Description: Days to regular opioid use from Timeline Followback
Time Frame: Up to Week 8 Post Discharge
Population: Patients admitted to detoxification or short term residential programs associated with CTN-0051 for OUD
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment As Usual
Number analyzed (Participants) | 211
days | 11.3 (11.58)

13. Primary Outcome: Days of Opioid Use
Description: Days of use up 8 weeks post discharge
Time Frame: Up to Week 8 Post Discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment As Usual
Number analyzed (Participants) | 211
days | 13.2 (16.7)

ADVERSE EVENTS:
Time Frame: 9 month
Description: For purposes of this study, only overdoses (whether hospitalized or not) and all deaths were collected. The relationship of adverse event was only collected for overdose events.
Groups:
- Treatment As Usual: Patients who were admitted to detoxification or short term residential programs associated with CTN-0051 with OUD.
Arm/Group | Treatment As Usual
All-Cause Mortality (participants affected / at risk) | 1/211
Serious Adverse Events (participants affected / at risk) | 7/211
Other Adverse Events (participants affected / at risk) | 8/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment As Usual (N=211)
Overdose (Respiratory, thoracic and mediastinal disorders) | 7 (7)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment As Usual (N=211)
Overdose (Respiratory, thoracic and mediastinal disorders) | 8 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT02730403/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT02730403/SAP_001.pdf